CLINICAL TRIAL: NCT04844541
Title: Prophylaxis and Treatment of COVID-19 - Adaptive Platform Trial
Brief Title: Prophylaxis and Treatment of COVID-19
Acronym: PROTECT-APT
Status: Completed | Type: Observational
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Joint Program Executive Office Chemical, Biological, Radiological, and Nuclear Defense Enabling Biotechnologies (Other Government)
Responsible Party: Sponsor
Other Study IDs: PC02
Record Dates: First submitted 2021-03-23; First posted 2021-04-14 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: COVID-19; Acute Respiratory Infection
Keywords: Point-of-Care Ultrasound; Physiological Monitoring; At Home Blood Collection; Patient-Centric Devices
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, Nasal mucus
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sub-population A Infected Cases: Symptomatic SARS-CoV-2 infected adults or adults meeting the ILI case definition (hospitalized and non-hospitalized)
- Sub-population B Contacts: Asymptomatic adult contacts of positive cases, defined as indoor exposure to the symptomatic case or cases within 6 feet (2 meters) for greater than or equal to 15 minutes over a 24-hour period without the use of personal protective equipment

SUMMARY:
An observation study evaluating physiologic responses and host biomarker expression patterns in early SARS-CoV-2 and acute respiratory infections (ARI) and among their close contacts.

DETAILED DESCRIPTION:
The aim of this observational study is to characterize the clinical, biological, virological, immunological, and pathological characteristics of ILI and SARS-CoV-2 infection in cases and their close contacts. The incorporation of novel technologies including self-specimen collection, symptom self-reporting, remote physiologic monitoring and virtual interaction with participants will enhance the capacity to conduct remote clinical trial activities. Inclusion of these remote and virtual elements into clinical trials augment the capacity to conduct much needed clinical research during times of resource strain such as a global pandemic. PROTECT-APT will be conducted as a multi-site study coordinated centrally by the Henry M Jackson Foundation for the Advancement of Military Medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Population A: Symptomatic SARS-CoV-2 or ILI Cases (hospitalized and non- hospitalized)

   1. Age ≥ 18 years old
   2. Presence of one or more of the following symptoms at enrollment:

      * Stuffy or runny nose
      * Hoarse voice
      * Sore throat
      * Difficulty breathing
      * Cough
      * Fatigue (Low energy or tiredness)
      * Muscle or body aches
      * Headache
      * Fever (documented temperature > 38°C [100.4°F]) or subjective fever
      * Chills or shivering
      * Feeling hot or feverish
      * Nausea
      * Vomiting
      * Diarrhea
      * Loss of smell
      * Loss of taste
   3. Positive molecular or antigen diagnostic test for SARS-CoV-2 at study enrollment or within ≤ 5 days prior to enrollment
   4. Symptom onset ≤ 5 days prior to enrollment

   OR
   1. Age ≥ 18 years old
   2. Meets the World Health Organization ILI case definition: An acute respiratory illness with a measured temperature of ≥ 38° C and cough, with onset within the past 10 days
2. Population B: SARS-CoV-2 or ILI Contacts

   1. Age ≥ 18 years old
   2. Asymptomatic contact of an individual with laboratory confirmed SARS-CoV-2 infection or an individual meeting the ILI case definition defined as:

      * Indoor exposure to the symptomatic case or cases within 6 feet (2 meters) for ≥ 15 minutes over a 24-hour period without the use of personal protective equipment
   3. For SARS-CoV-2 contacts: Negative screening SARS-CoV-2 molecular or antigen diagnostic test performed at screening or within ≤ 24 hours of enrollment
   4. Exposure and enrollment within 6 days or less from when the symptomatic, confirmed SARS-CoV-2 or ILI case first had symptoms

Exclusion Criteria:

1. Population A: Adults seeking care or testing for SARS-CoV-2 or ILI

   a. Laboratory confirmed SARS-CoV-2 infection 6 to 90 days prior to enrollment
2. Population B: Adult contacts of SARS-CoV-2 or ILI infected individuals

   1. Symptoms attributed to COVID-19 or ILI as assessed by a medical provider
   2. Positive molecular or antigen test for SARS-CoV-2 from any upper respiratory specimen within 90 days prior to enrollment
   3. SARS-CoV-2 vaccination within 90 days prior to enrollment EXCEPT if severely immunocompromised or a known vaccine non-responder

      * Severely immunocompromised or a known vaccine non-responder defined as: solid organ or stem cell recipient, B cell leukemia, receiving B cell depletion therapy (e.g., rituximab), agammaglobulinemia, or negative serology ≥ 2 weeks after vaccination with two doses of a vaccine
   4. Positive PCR test for acute respiratory infection including but not limited to influenza, RSV, adenovirus, parainfluenza virus, rhinovirus, metapneumovirus, Bordatella Pertussis, Chlamydia Pneumonia, coronavirus (other than SARS-CoV-2), mycoplasma within 7 days of enrollment
   5. Hospital admission at the time of enrollment

      * Hospitalization will be defined as requiring medical care not available in an outpatient setting for greater than 24 hours.
      * Hospitalization for isolation or quarantine requirements or for social reasons will NOT constitute an exclusion criterion

For Both populations:

1. Absence of informed consent
2. Individuals who the study investigators believe are unable to comply with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population A. Infected Cases:
  Symptomatic SARS-CoV-2 infected adults or Adults meeting the ILI case definition
  Population B. Contacts:
  Asymptomatic adult contacts of positive cases, defined as indoor exposure to they symptomatic case or cases within 6 feet (2 meters) for greater than or equal to fifteen minutes over a 24-hour period without the use of personal protective equipment
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Time-weighted average change in symptom score | 12 Weeks
  Describe the clinical characteristics of ILI and SARS-CoV-2 in the target populations
Number of days with symptoms | 12 Weeks
  Describe the clinical characteristics of ILI and SARS-CoV-2 in the target populations

SECONDARY OUTCOMES:
Proportion of ILI and SARS-CoV-2 infected adults seeking non-scheduled care for ILI and SARS-CoV-2 | 12 Weeks
  Describe the biological, virological, immunological, and pathological characteristics of ILI and SARS-CoV-2 in the target populations
Time to clearance of SARS-CoV-2 in upper respiratory specimens of ILI and SARS-CoV-2 infected adults | 12 Weeks
  Describe the biological, virological, immunological, and pathological characteristics of ILI and SARS-CoV-2 in the target populations
Rate of change from the SARS-CoV-2 maximal viral load in ILI and SARS-CoV-2 infected adults | 28 Days
  Describe the biological, virological, immunological, and pathological characteristics of ILI and SARS-CoV-2 in the target populations
Proportion of lab confirmed infections (e.g., SARS-CoV-2, influenza, coronavirus except SARS-CoV-2, RSV, parainfluenza, adenovirus, rhinovirus, metapneumovirus, B. Pertussis, C. Pneumonia, mycoplasmas) in uninfected adult contacts | 12 Weeks
  Describe the biological, virological, immunological, and pathological characteristics of ILI and SARS-CoV-2 in the target populations
Time-weighted average change from baseline viral load in SARS-CoV-2 uninfected adult contacts who become infected | 14 Days
  Describe the biological, virological, immunological, and pathological characteristics of ILI and SARS-CoV-2 in the target populations
Change in modified ordinal outcome scale | 12 Weeks
  Describe the biological, virological, immunological, and pathological characteristics of ILI and SARS-CoV-2 in the target populations
Time-weighted average change in lung fields with B lines using point of care lung ultrasound | 12 Weeks
  Describe the biological, virological, immunological, and pathological characteristics of ILI and SARS-CoV-2 in the target populations
Change in SARS-CoV-2 IgM, IgG, and neutralizing antibodies from baseline | 12 Weeks
  Describe the biological, virological, immunological, and pathological characteristics of ILI and SARS-CoV-2 in the target populations

OTHER OUTCOMES:
Host gene expression levels that predict ILI or SARS-CoV-2 progression | 12 Weeks
  Identify baseline and longitudinal host and pathogen factors predictive of progression to guide clinical triage and treatment decisions
Host protein biomarkers that predict ILI or SARS-CoV-2 progression | 12 Weeks
  Identify baseline and longitudinal host and pathogen factors predictive of progression to guide clinical triage and treatment decisions
Immunophenotypes that predict ILI or SARS-CoV-2 progression | 12 Weeks
  Identify baseline and longitudinal host and pathogen factors predictive of progression to guide clinical triage and treatment decisions
Physiologic markers that predict ILI or SARS-CoV-2 progression | 12 Weeks
  Identify baseline and longitudinal host and pathogen factors predictive of progression to guide clinical triage and treatment decisions

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Clark, PhD, Study Chair — Henry M. Jackson Foundation for the Advancement of Military Medicine
Locations (3):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Duke Global Health Institute, Durham, North Carolina
- Royal Thai Army Clinical Research Center (RTA CRC)/Royal Thai Army-Armed Forces Research Institute of Medical Sciences (RTA-AFRIMS)/Phramongkutklao Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided